CLINICAL TRIAL: NCT02771509
Title: A Multicenter, Prospective, Parallel-Group, Double-Blind, Randomized, Placebo-Controlled, Phase 2 Study of ANG-3777 to Assess the Safety and Efficacy of BB3 in Patients Developing Acute Kidney Injury After Cardiac Surgery
Brief Title: Study to Prevent Acute Kidney Injury After Cardiac Surgery Involving Cardiopulmonary Bypass
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Angion Biomedica Corp (Industry)
Collaborators: Everest Clinical Research (Unknown); CTI Clinical Trial and Consulting Services (Other); Clinical Accelerator (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 002-15
Record Dates: First submitted 2016-04-18; First posted 2016-05-13 (Estimated); Last update posted 2021-07-15 (Actual); Status verified 2021-07

CONDITIONS: Acute Kidney Injury
Keywords: CPB; Cardiac Surgery; Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury | interventions — terevalefim; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ANG-3777 (Active Comparator): Study drug will be administered for a total of 4 daily intravenous (IV) infusions. The first post-operative dose MUST be started within 4 hours of completing CPB. The second dose will be administered 24 ± 2 hours after completing CPB, and the third and fourth doses will be administered 24 ± 2 hours after each previous dose. Duration of administration is 30 minutes.
  Interventions: Drug: ANG-3777
- Normal Saline (Placebo Comparator): The placebo will be administered for a total of 4 daily intravenous (IV) infusions. The first post-operative dose MUST be started within 4 hours of completing CPB. The second dose will be administered 24 ± 2 hours after completing CPB, and the third and fourth doses will be administered 24 ± 2 hours after each previous dose. Duration of administration is 30 minutes.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ANG-3777 — 6 mg/mL BB3, IV, 4 days in a row, first dose must be within 4 hours after surgery, the next three doses will be approx. 24 hours after the last dose
  Other Names: Hepatocyte growth factor mimetic
  Arms: ANG-3777
Drug: Placebo — Normal saline
  Other Names: Normal Saline
  Arms: Normal Saline

SUMMARY:
The objective of the study is to assess the safety and efficacy of ANG-3777 in preventing AKI compared to placebo when administered to patients at risk for developing acute kidney injury (AKI) following cardiac surgical procedures involving cardiopulmonary bypass (CPB).

ELIGIBILITY:
Inclusion Criteria:

1. Patient is either male or female ≥ 18 years.
2. Patient has provided written informed consent, and is willing and able to comply with the requirements of the study protocol, including screening procedures.
3. Patient must be scheduled for and undergo a non-emergent cardiac surgical procedure involving CPB. Eligible procedures include:

   1. Coronary artery bypass graft (CABG) alone
   2. Aortic valve replacement or repair alone, with or without aortic root repair
   3. Mitral, tricuspid, or pulmonic valve replacement or repair alone
   4. Combined replacement of several cardiac valves
   5. CABG with aortic, mitral, tricuspid, or pulmonic valve replacement or repair
   6. CABG with combined cardiac valve replacement or repair.
4. Patient must have the following risk factor(s) for AKI prior to surgery:

   1. Estimated glomerular filtration rate (eGFR) of ≥ 20 and < 30 ml/min/1.73m2, or
   2. eGFR ≥ 30 and < 60 mL/min/1.73m2 and ONE of the following Additional Risk Factors (other than age ≥ 75 years), or
   3. eGFR ≥ 60 ml/min/1.73m2 and TWO of the following Additional Risk Factors

   eGFR will be calculated using the abbreviated MDRD equation (MDRD-4, often referred to as the Levey equation): eGFR = 186.3 x sCr-1.154 x Age-0.203 x [0.742 if Female] x [1.212 if Black]

   Additional Risk Factors:
   * Combined valve and coronary surgery
   * Previous cardiac surgery with sternotomy
   * Left ventricular ejection fraction (LVEF) < 35% by invasive or noninvasive diagnostic cardiac imaging within 90 days prior to surgery
   * Diabetes mellitus requiring insulin treatment
   * Non-insulin-requiring diabetes with documented presence of at least moderate (+2 or > 100 mg/dL) proteinuria on urine analysis (medical history or dipstick)
   * Documented NYHA Class III or IV within 1 year prior to index surgery
   * Age ≥ 75 years can be considered an Additional Risk Factor only for patients with eGFR ≥ 60 ml/min/1.73m2.
5. Patient must have presented for surgery without prior evidence of active renal injury defined as no acute rise in sCr > 0.3 mg/dL or no 50% increase in sCr between the time of Screening and pre-surgery.
6. Patient's body mass index (BMI) < 40 at Screening.

Exclusion Criteria:

1. Patient has eGFR < 20 mL/min/1.73 m2 within 48 hours pre-surgery as measured by MDRD 4.
2. Patient has ongoing sepsis or partially treated infection. Sepsis is defined as the presence of a confirmed pathogen, along with fever or hypoperfusion (i.e., acidosis and new onset elevation of liver function tests) or hypotension requiring pressor use prior to surgery.
3. Currently active infection requiring antibiotic treatment.
4. Patient who has an active (requiring treatment) malignancy or history within 5 years prior to enrollment in the study, of solid, metastatic or hematologic malignancy with the exception of basal or squamous cell carcinoma of the skin that has been removed.
5. Administration of iodinated contrast material within 24 hours prior to cardiac surgery.
6. Patients diagnosed with AKI as defined by KDIGO criteria within 48 hours prior to surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 275 (Actual)
Dates: Start 2017-02-24 (Actual); Primary Completion 2021-08 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
The mean AUC of the percent increase in serum creatinine above baseline | starting from 24 hr after the end of CPB through Day 6

CONTACTS AND LOCATIONS:
Overall Officials: John Neylan, MD, Study Director — Angion Biomedica
Locations (40):
- United States (23):
  - University of Southern California, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Stanford University Medical Center, Palo Alto, California
  - California Institute of Renal Reseach, San Diego, California
  - Yale University School of Medicine, New Haven, Connecticut
  - Fleming Island Center for Clinical Research, Fleming Island, Florida
  - UF Health at Unviersity of Florida, Gainesville, Florida
  - River City Clinical Research, Jacksonville, Florida
  - Indiana Ohio Heart, Fort Wayne, Indiana
  - University of Maryland Medical Center, Baltimore, Maryland
  - Suburban Hospital, Bethesda, Maryland
  - MidMichigan Medical Center Midland, Midland, Michigan
  - Cardiac & Vascular Research Center of Northern Michigan, Petoskey, Michigan
  - Bryan Heart, Lincoln, Nebraska
  - Columbia University Medical Center, New York, New York
  - Duke University, Durham, North Carolina
  - Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - TriHealth, Cincinnati, Ohio
  - Cleveland Clinic Fairview, Cleveland, Ohio
  - Ohio State Wexner Medical Center, Columbus, Ohio
  - Baylor Jack and Jane Hamilton Heart and Vascular center- Soltero Cardiovascular Research Center, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - University of Virginia Health System, Charlottesville, Virginia
- Brazil (5):
  - Faculdade de Medicina da UNESP Campus de Botucatu, Botucatu
  - Instituto de Cardiologia do Rio Grande do Sul / Fundação Universitária de Cardiologia (IC - FUC), Porto Alegre
  - Hospital das Clínicas da Faculdade de Medicina de Ribeirão Preto da Universidade de São Paulo (HCFMRP), Ribeirão Preto
  - Fundação Faculdade Regional de Medicina de São José do Rio Preto, São José do Rio Preto
  - Instituto do Coração do Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo (InCor - HCFMUSP), São Paulo
- Canada (6):
  - St. John Regional Hospital, Saint John, New Brunswick
  - London Health Sciences Center, London, Ontario
  - Saint Michael's Hospital, Toronto, Ontario
  - CHUM - Hôtel Dieu, Montreal, Quebec
  - MUHC - Royal Victoria Hospital, Montreal, Quebec
  - Institut Universitaire de Cardiologie et de Pneumologie de Québec, Québec
- Georgia (6):
  - Israeli-Georgian Medical Research Clinic Helsicore, Tbilisi
  - New Hospitals LTD, Tbilisi
  - Bokhua Memorial Cardiovascular Center, Tbilisi
  - Jerarsi JSC, Tbilisi
  - Tbilisi Heart Center, Tbilisi
  - Acad. G. Chapidze Emergency Cardiology Center, Tbilisi